CLINICAL TRIAL: NCT02959879
Title: Resectable Pancreatic Adenocarcinoma Neo-Adjuvant FOLF(IRIN)OX-based CHEmotherapy - A Multicenter, Randomised Phase II Trial (PANACHE01-PRODIGE48 Study)
Brief Title: Neo-adjuvant FOLF(IRIN)OX for Resectable Pancreatic Adenocarcinoma
Acronym: PANACHE01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: UNICANCER (Other); Federation Francophone de Cancerologie Digestive (Other); Federation of Research in Surgery (FRENCH) (Other); GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/0210/HP
Record Dates: First submitted 2016-11-03; First posted 2016-11-09 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2018-04

CONDITIONS: Resectable Pancreatic Duct Adenocarcinoma
Keywords: FOLFOX; FOLFIRINOX
MeSH Terms: interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FOLFOX neoadjuvant chemotherapy (Experimental): 4 cycles of FOLFOX neoadjuvant chemotherapy are administrated to patient. Curative surgery for resectable pancreatic duct adenocarcinoma will be done after neoadjuvant chemotherapy. 8 cycles of adjuvant chemotherapy are administrated following the surgery
  Interventions: Drug: FOLFOX neoadjuvant chemotherapy; Procedure: curative surgery for resectable pancreatic duct adenocarcinoma; Drug: adjuvant chemotherapy
- FOLFIRINOX neoadjuvant chemotherapy (Experimental): 4 cycles of FOLFIRINOX neoadjuvant chemotherapy are administrated to patient. Curative surgery for resectable pancreatic duct adenocarcinoma will be done after neoadjuvant chemotherapy. 8 cycles of adjuvant chemotherapy are administrated following the surgery
  Interventions: Drug: FOLFIRINOX neoadjuvant chemotherapy; Procedure: curative surgery for resectable pancreatic duct adenocarcinoma; Drug: adjuvant chemotherapy
- standard adjuvant chemotherapy (Active Comparator): Curative surgery for resectable pancreatic duct adenocarcinoma will be done after randomization.
  12 cycles of standard adjuvant chemotherapy are administrated following the surgery
  Interventions: Procedure: curative surgery for resectable pancreatic duct adenocarcinoma; Drug: Standard adjuvant chemotherapy

INTERVENTIONS:
Drug: FOLFOX neoadjuvant chemotherapy — 4 cycles of FOLFOX neoadjuvant chemotherapy are administrated to patient
  Arms: FOLFOX neoadjuvant chemotherapy
Drug: FOLFIRINOX neoadjuvant chemotherapy — 4 cycles of FOLFIRINOX neoadjuvant chemotherapy are administrated to patient
  Arms: FOLFIRINOX neoadjuvant chemotherapy
Procedure: curative surgery for resectable pancreatic duct adenocarcinoma — curative surgery for resectable pancreatic duct adenocarcinoma
Drug: Standard adjuvant chemotherapy — 12 cycles of standard adjuvant chemotherapy are administrated
  Arms: standard adjuvant chemotherapy
Drug: adjuvant chemotherapy — 8 cycles of standard adjuvant chemotherapy are administrated
  Arms: FOLFIRINOX neoadjuvant chemotherapy; FOLFOX neoadjuvant chemotherapy

SUMMARY:
In patients with resectable pancreatic duct adenocarcinoma (PDAC), curative surgery followed by adjuvant chemotherapy is currently the standard of care. However, the long-term results are still poor, with median disease-free and overall survival of 14 months and 23 months. The corresponding 5-year overall survival rate is 20%.

Chemotherapy before surgery (neoadjuvant chemotherapy) allows identification of patients with rapidly progressive metastatic disease at time of preoperative restaging (surgery is then avoided in these patients), and may increase the rate of free margin resection (R0) and reduce the risk of local recurrence.

Even though single-agent gemcitabine and 5-FU have been validated in adjuvant and metastatic settings, the objective response was low (at around 10%), whereas combination chemotherapy exceeds a response rate of 30% in advanced disease. In metastatic PDAC, palliative FOLFIRINOX chemotherapy has been demonstrated to be effective (in terms of response rates and progression-free survival) and well tolerated. Interestingly, the response rate is increased by using more than two chemotherapeutic agents in advanced pancreatic cancer, justifying the use of an alternative neoadjuvant FOLFOX-based chemotherapy arm.

PANACHE-01 is an open, non-comparative, randomised, multicentre Phase II study designed to assess the safety and efficacy of two modes of neo-adjuvant chemotherapy (FOLFIRINOX & FOLFOX) relative to the current reference treatment (surgery and then adjuvant chemotherapy) for resectable PDAC.

Patients with immediately resectable PDAC (definition based on the NCCN's (American National Comprehensive Cancer Network 2014) latest guidelines) will be randomised to either pancreatectomy and adjuvant chemotherapy or 4 cycles of neoadjuvant chemotherapy with either FOLFOX or FOLFIRINOX. The patients in the neoadjuvant chemotherapy arms will receive postoperative chemotherapy for 4 months (8 cycles).

ELIGIBILITY:
Inclusion Criteria:

* Histology-proven, adenocarcinoma of the pancreas.
* Resectable adenocarcinoma (according to the NCCN classification 2014): absence of distant organ or distal lymph node metastases, absence of evidence of superior mesenteric vein (SMV) and portal vein distortion, tumour thrombus, or venous encasement, the existence of clear fat planes around the celiac axis, hepatic artery and superior mesenteric artery (SMA). Resectability is evaluated on arterial-phase and portal-phase IV contrast-enhanced multislice CT-scan of the pancreas (slice thickness: 2.5 mm), as evaluated in a multidisciplinary staff meeting including at least one radiologist and one expert surgeon.
* No prior chemotherapy.
* Age 18 years or over.
* Ability to understand and willingness to consent to formal requirements for study participation
* Provision of written informed consent prior to any study-specific screening procedures.

Exclusion Criteria:

* PDAC defined as "borderline", locally advanced, non-resectable or metastatic.
* Prior cancer therapy for PDAC
* Surgical or anaesthesiological contra-indications: non-controlled congestive heart failure - non-treated angina - recent myocardial infarction (in the previous year) - non-controlled arterial hypertension (SBP >160 mm or DBP > 100 mm, despite optimal drug treatment), long QT, major non-controlled infection, severe liver failure.
* Any medical, psychological or social situation that (in the investigator's opinion) could limit (i) the patient's compliance with the protocol or (ii) the ability to obtain or interpret data.
* Pregnant or breastfeeding women and women of child-bearing age not using effective means of contraception.
* History or current evidence on physical examination of central nervous system disease or peripheral neuropathy ≥ grade 1, according to according to Common Terminology Criteria for Adverse Events (CTCAE) v.4.0.
* Known hypersensitivity reaction to any of the components of study treatments.
* Pregnancy (the absence of which must be confirmed in a ß-hCG test) or breast-feeding.
* Any significant disease which, in the investigator's opinion, would exclude the patient from the study.
* Patients having been included in a clinical trial within the previous 4 weeks or participating in another trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Number of patients alive | 12 months
  Number of patients alive is evaluated 12 months after the surgery
Number of patients who achieved the complete chemotherapy treatment sequences | 12 months
  The number of patients who achieved the complete chemotherapy treatment sequences is evaluated 12 months after the surgery

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | through end of treatment, an average of 12 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Number of post-operative complications | 1 month after surgery
  Evaluation of post-operative complications is assessed using Dindo Clavien classification
Number of patients alive and without recurrence | 36 months
  Number of patients alive is evaluated 36 months after the surgery
Number of accomplished R0 resection surgery | Surgery day
  Number of accomplished R0 resection surgery is evaluated by pathologists
Evaluation of quality of life | 4 weeks after the end of chemotherapy treatment
  Evaluation of quality of life is done using EORTC QLQ C30
Evaluation of quality of life | 4 weeks after the end of chemotherapy treatment
  Evaluation of quality of life is done using EORTC QLQ-PAN26

CONTACTS AND LOCATIONS:
Overall Officials: Lilian SCHWARZ, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schwarz L, Bachet JB, Meurisse A, Bouche O, Assenat E, Piessen G, Hammel P, Regenet N, Taieb J, Turrini O, Paye F, Turpin A, Souche FR, Laurent C, Kianmanesh R, Michel P, Vernerey D, Mabrut JY, Turco C, Truant S, Sa Cunha A; PANACHE01-FRENCH08-PRODIGE48 Investigators. Neoadjuvant FOLF(IRIN)OX Chemotherapy for Resectable Pancreatic Adenocarcinoma: A Multicenter Randomized Noncomparative Phase II Trial (PANACHE01 FRENCH08 PRODIGE48 study). J Clin Oncol. 2025 Jun 10;43(17):1984-1996. doi: 10.1200/JCO-24-01378. Epub 2025 Apr 4. PMID 40184561
- [Derived] Schwarz L, Vernerey D, Bachet JB, Tuech JJ, Portales F, Michel P, Cunha AS. Resectable pancreatic adenocarcinoma neo-adjuvant FOLF(IRIN)OX-based chemotherapy - a multicenter, non-comparative, randomized, phase II trial (PANACHE01-PRODIGE48 study). BMC Cancer. 2018 Jul 24;18(1):762. doi: 10.1186/s12885-018-4663-4. PMID 30041614